CLINICAL TRIAL: NCT03457376
Title: Correlation of the Hand Grip Force With Maximum Inspiratory and Maximum Expiratory Pressure, in Critical Ill Patients
Status: Completed | Type: Observational
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Konstantinos Grigoriadis, PT, MSc, PhD, Attikon Hospital
Other Study IDs: EBD2877/06-12-2017
Record Dates: First submitted 2018-03-01; First posted 2018-03-07 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Intensive Care Unit Syndrome
MeSH Terms: interventions — Maximal Respiratory Pressures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Hand Grip Force — Hand Grip Force
Diagnostic Test: Maximal Inspiratory Pressure — Maximal Inspiratory Pressure
Diagnostic Test: Maximal Expiratory Pressure — Maximal Expiratory Pressure

SUMMARY:
This study aimed to examine the relationship between Hand Grip Force (HGF), Maximum Inspiratory Pressure (PImax) and Maximum Expiratory Pressure (PEmax) in ICU tracheostomized patients. METHODS: All patients underwent assessment of PImax and PEmax by a membrane-type manometer, and for the measure of HGF an hydraulic hand dynamometer

DETAILED DESCRIPTION:
Design of the study This is a random retrospective observational study concerned the period from 5/2017 to 1/2018. The study was conducted for patients of the 2nd General University Intensive Care Unit, of Attikon University General Hospital. The data studied as a sample are derived from file records of adult male and female ICU patients.

The inclusion - exclusion criteria

* Adult ICU patients
* Stable haemodynamic
* Who were able to perform commands from breathing exercises in their hospitals in the ICU (Glasgow Comma Scale 15) good communication and level of consciousness in order to be able to execute orders
* Have integers limbs
* Were tracheostomy (measurements in this case result from a special adapter in the tracheostomy that ensures minimization of losses)
* Their stay in the ICU should have been more than 11 days (the incidence of ICU muscle weakness occurs after 7 days of hospitalization19).
* In order to ensure the randomness of the sample, records of patients who were only hospitalized on an even bed number.
* All requirements for patient recruitment were solely for the day of the study
* They should not suffer from any neurological syndrome (central or peripheral type) other than the ICU acquired weakness, or even craniocerebral injury that could have an effect on the peripheral muscle strength.
* Without drugs that could affect perception or muscle tone Measurements Τhe blindness of the study was ensured because both evaluators and patients don't know were participating in a study. The data from records on patient files related to the following: PEmax, PImax, HG, Age, Weight, Height, points in Glasgow Coma Scale, creatinine, use of inotrope drugs, partial pressure of oxygen (PaO2), platelets, bilirubin, oxygen supply (FiO2), cause of admission and day of hospitalization in the ICU. The last eight values are taken to calculate the SOFA to determine the severity of the condition of these patients. Finally, due to the use of historical data from the patient file, it was not considered necessary to obtain a paper consensus.

Statistical analysis Descriptive statistics are presented as means ± SD, medians and interquartile ranges, or percentages when appropriate. The Shapiro -Wilk test was used to determine whether the variables of interest followed a normal distribution. For the calculation of the correlation between parametric variables Pearson's correlation test was used, and for the calculation of the correlation between non parametric variables Spearman's rho was used. Rho coefficient correlation of <0.20 is considered to indicate very weak correlation, 0.21-0.40 indicates weak correlation, 0.41- 0.60 indicates moderate correlation and 0.61-0.80 indicates strong correlation. Finally a linear regression analysis was run to predict HGF from PEmax.

ELIGIBILITY:
Inclusion Criteria:

* Adult ICU patients
* Stable haemodynamic
* Who were able to perform commands from breathing exercises in their hospitals in the ICU (Glasgow Comma Scale 15) good communication and level of consciousness in order to be able to execute orders
* Have integers limbs
* Were tracheostomy (measurements in this case result from a special adapter in the tracheostomy that ensures minimization of losses)
* Their stay in the ICU should have been more than 11 days (the incidence of ICU muscle weakness occurs after 7 days of hospitalization19).
* In order to ensure the randomness of the sample, records of patients who were only hospitalized on an even bed number.
* All requirements for patient recruitment were solely for the day of the study

Exclusion Criteria:

* They should not suffer from any neurological syndrome (central or peripheral type) other than the ICU acquired weakness, or even craniocerebral injury that could have an effect on the peripheral muscle strength.
* Without drugs that could affect perception or muscle tone

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ICU patients Tracheostomized Age, mean ± SD; median (IQR) y 67.2 ± 13.6; 74 (59.6-74.7) Male subjects 12 Weight, mean ± SD; median (IQR) kg 80 ± 15.2; 75 (71.5-88.4) Height, mean ± SD; median (IQR) cm 169 ± 9; 170 (164-174) PImax, mean ± SD; median (IQR) cm H2O 36.4 ± 12.1; 35 (29.6-43.1) PEmax, mean ± SD; median (IQR) cm H2O 40 ± 11.5; 40 (33.9-46.8) HGF, mean ± SD; median (IQR) kg 10.8 ± 7.9; 10 (6.3-15.2) BMI, mean ± SD; median (IQR) kg/m2 27.8 ± 5.4; 27.8 (24.7-30.8) ICU day of Hospitalization 20.6 ± 8.4; 20 (15.9-25.3) SOFA score 3.5 ± 1.5; 3 (2.6-4.3)
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Correlation PImax and Hand Grip Force | 9 Mοnths
  Correlation PImax and Hand Grip Force
Correlation PEmax and Hand Grip Force | 9 Months
  Correlation PEmax and Hand Grip Force

CONTACTS AND LOCATIONS:
Overall Officials: Apostolos Armaganidis, Professor, Study Director — Attikon University Hospital, ICU
Locations (2):
- Greece (2):
  - Attikon University Hospital, Athens, Attica
  - Grigoriadis Konstantinos, Athens, Attica

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Jonghe B, Bastuji-Garin S, Durand MC, Malissin I, Rodrigues P, Cerf C, Outin H, Sharshar T; Groupe de Reflexion et d'Etude des Neuromyopathies en Reanimation. Respiratory weakness is associated with limb weakness and delayed weaning in critical illness. Crit Care Med. 2007 Sep;35(9):2007-15. doi: 10.1097/01.ccm.0000281450.01881.d8. PMID 17855814
- [Background] Bahat G, Tufan A, Ozkaya H, Tufan F, Akpinar TS, Akin S, Bahat Z, Kaya Z, Kiyan E, Erten N, Karan MA. Relation between hand grip strength, respiratory muscle strength and spirometric measures in male nursing home residents. Aging Male. 2014 Sep;17(3):136-40. doi: 10.3109/13685538.2014.936001. Epub 2014 Jul 4. PMID 24993454
- [Result] Volianitis S, McConnell AK, Jones DA. Assessment of maximum inspiratory pressure. Prior submaximal respiratory muscle activity ('warm-up') enhances maximum inspiratory activity and attenuates the learning effect of repeated measurement. Respiration. 2001;68(1):22-7. doi: 10.1159/000050458. PMID 11223726
- [Result] Steier J, Kaul S, Seymour J, Jolley C, Rafferty G, Man W, Luo YM, Roughton M, Polkey MI, Moxham J. The value of multiple tests of respiratory muscle strength. Thorax. 2007 Nov;62(11):975-80. doi: 10.1136/thx.2006.072884. Epub 2007 Jun 8. PMID 17557772
- [Result] Shin HI, Kim DK, Seo KM, Kang SH, Lee SY, Son S. Relation Between Respiratory Muscle Strength and Skeletal Muscle Mass and Hand Grip Strength in the Healthy Elderly. Ann Rehabil Med. 2017 Aug;41(4):686-692. doi: 10.5535/arm.2017.41.4.686. Epub 2017 Aug 31. PMID 28971054
- [Result] Efstathiou ID, Mavrou IP, Grigoriadis KE. Correlation Between Maximum Inspiratory Pressure and Hand-Grip Force in Healthy Young and Middle-Age Individuals. Respir Care. 2016 Jul;61(7):925-9. doi: 10.4187/respcare.04319. Epub 2016 Apr 19. PMID 27094394
- [Derived] Grigoriadis K, Efstathiou I, Dimitriadis Z, Konstantopoulou G, Grigoriadou A, Vasileiadis G, Micha M, Tsagaris I, Armaganidis A. Handgrip Force and Maximum Inspiratory and Expiratory Pressures in Critically Ill Patients With a Tracheostomy. Am J Crit Care. 2021 Mar 1;30(2):e48-e53. doi: 10.4037/ajcc2021248. PMID 33644812